CLINICAL TRIAL: NCT02864342
Title: A Randomized Clinical Study to Assess the Impact of Symbicort® pMDI Medication Reminders on Adherence in COPD Patients
Brief Title: Adherence Study in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: D589CL00003
Record Dates: First submitted 2016-07-26; First posted 2016-08-12 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD
Keywords: chronic obstructive pulmonary disease; COPD; Respiratory; adherence; medication reminders
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BreatheMate device and application (Active Comparator): BreatheMate Bluetooth device that attaches to Symbicort pressurized Metered Dose Inhaler (pMDI) and cell phone with application that sends medication and refill reminders and reminders to complete a COPD questionnaire
  Interventions: Device: Arm 1: BreatheMate device with application
- BreatheMate device without application (Placebo Comparator): BreatheMate Bluetooth device that attaches to Symbicort pressurized Metered Dose Inhaler (pMDI) and cell phone without any reminders or alerts.
  Interventions: Device: Arm 2: BreatheMate device without application

INTERVENTIONS:
Device: Arm 1: BreatheMate device with application — The service known as 'BreatheMate' is a patient support tool that monitors daily Symbicort inhaler use. The BreatheMate service includes a bluetooth monitoring device that is attached to subjects' Symbicort pMDI inhaler which automatically detects and logs their maintenance medication use. Subjects will receive audio-visual daily reminders (beeps and flashes) on the BreatheMate Bluetooth device. The bluetooth device transmits this data to a cellular phone that is provided to all subjects in the study. Subjects in the intervention group will also receive audio-visual alerts (beeps, flashes) from the bluetooth device to take their medication.
  Arms: BreatheMate device and application
Device: Arm 2: BreatheMate device without application — The service known as 'BreatheMate' is a patient support tool that monitors daily Symbicort inhaler use. The BreatheMate service includes a bluetooth monitoring device that is attached to subjects' Symbicort pMDI inhaler which automatically detects and logs their maintenance medication use. The functionality of audio-visual daily reminders (beeps and flashes) is deactivated for this control group.
  The BreatheMate service also includes a cellular phone that will display whether the Bluetooth monitoring device is paired and communicating with the cellular phone. The Bluetooth device will transmit data regarding medication usage to the cellular phone.
  Arms: BreatheMate device without application

SUMMARY:
A randomized clinical study to assess the impact of Symbicort® pMDI medication reminders on adherence in COPD patients

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common disease with substantial associated morbidity and mortality. COPD is the third leading cause of death in the US and claimed 133,965 US lives in 2009. In 2011 12.7 million US adults were estimated to have COPD. However, approximately 24 million US adults have evidence of impaired lung function, indicating an under diagnosis of COPD. COPD also has a potentially harmful economic impact. In 2010, COPD resulted in over 10 million office visits, nearly 1.5 million emergency department visits, 700,000 hospitalizations, and 133,575 deaths in the US. In 2010, US total medical treatment costs attributed solely to COPD (i.e., excluding comorbidities) were estimated to be $32.1 billion with an additional $3.9 billion in COPD costs resulting from worker absenteeism. Even in industrialized countries such as the US, where anti-smoking initiatives have been relatively successful, the legacy of past smoking behavior in aging populations ensures that the COPD burden will unavoidably continue to climb over the next 20 to 30 years. Adherence rates for inhaled combination therapy is poor (average 3.9 refills per year). COPD patients with lower adherence tend to have higher overall healthcare costs, as demonstrated in a 24 month study of 33,816 patients in the US, which found: Patients continuing therapy had lower costs of care by $3764 compared with patients who had ceased to take their maintenance therapy. COPD patients with higher adherence to prescribed regimens experienced fewer hospitalizations and lower Medicare costs (-$2185) than those who exhibited lower adherence behaviors. Given the poor adherence with inhaled combination therapy seen in patients with COPD, and associated morbidity/mortality and economic costs, the present study is being conducted to see if medication reminders can be used to improve adherence in this population.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfil the following criteria:

* Signed informed consent at Visit 1 prior to any study specific procedures
* Outpatient adults 40 years and older
* A diagnosis of COPD confirmed by a post-bronchodilator Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) <0.70 at some point in the past 3 years.
* Moderate to Very Severe COPD as defined by a post-bronchodilator FEV1 <80% of predicted on most recent spirometry.
* Had been on an ICS/LABA combination therapy of a brand and dose approved forCOPD, for at least 3 months prior to screening.
* Current or previous smoker with a smoking history equivalent to 10 or more pack years (1 pack year = 20 cigarettes smoked per day for 1 year).
* Willing to discontinue all medications containing both a LABA and an ICS and to begin Symbicort 160/4.5 μg, 2 inhalations bid.
* Must be willing to make a return visit, and complete all study assessments for the duration of study.
* Life expectancy >12 months.
* Must be willing to comply with all study procedures including being able to remove and attach device to the inhaler.
* Must be able and willing to read and write/respond using the electronic device provided.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Previous randomization in the present study.
* Patients who have been randomized in a clinical study and received an investigational product within 30 days of Visit 1 (participation is defined as the completion of a treatment related visit).
* Current diagnosis of asthma.
* Known history of drug or alcohol abuse which, in the opinion of the Investigator, may interfere with subject's ability to participate or comply with the study.
* An acute exacerbation of COPD that required hospitalization or emergency room visit or treatment with systemic steroids and/or antibiotics during the 28 days before Visit 1. Patients who had a COPD exacerbation within 28 days of Visit 1 can be re-screened once. Re-screening can occur no earlier than 28 days from the last dose of systemic steroids and/or antibiotics and/or hospitalization, whichever is later.
* Enrolled patients that have a COPD exacerbation during the run-in period, defined as worsening symptoms which in the judgment of the Investigator requires treatment with systemic steroids and/or antibiotics and/or hospitalization. Patients who had a COPD exacerbation during the run-in period can be re-screened once. Re-screening can occur no earlier than 28 days from the last dose of systemic steroid and/or antibiotics and/or hospitalization, whichever is later.
* Any hospital admissions due to ischemic heart disease or heart failure within 3 months of study enrollment.
* Any significant disease or disorder (e.g., gastrointestinal, liver, renal, neurologic, musculoskeletal, endocrine, metabolic, infectious, psychiatric, major physical impairment) which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study.
* History of lung or upper airway cancer and any other malignancy not in remission for 5 years or more, except for patients who have had basal cell carcinoma, or in situ carcinoma of the cervix provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained.
* Use or planned use of systemic corticosteroids as a maintenance treatment (defined as daily or every other day treatment for 21 or more days) for inflammatory or immunologic conditions unrelated to their COPD.
* Planned hospitalization or surgical procedure requiring inpatient stay during the study.
* Pregnancy, breast-feeding or planned pregnancy during the study; fertile women not using acceptable contraceptive measures, as judged by the Investigator. Female subjects who are not post-menopausal or surgically sterile must have a negative urine pregnancy test (urine dipstick test only) prior to randomization and must comply with contraceptive methods.
* Any clinically relevant abnormal findings in physical examination or vital signs, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study.
* Known or suspected hypersensitivity to the study therapy (Symbicort).
* Patients who are unable or unwilling to use mobile communication devices, or patients who plan to be away from home for a significant part of the study without access to cellular connectivity are excluded because of the challenges of collecting data and providing information to these patients who are unable to use the service.
* Patients with thoracic surgery within 6 months of Visit 1.
* Patients who have received a lung transplant or are currently active on the lung transplant waiting list.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Research Site, Clearwater, Florida
  - Research Site, Tampa, Florida
  - Research Site, Marlton, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Spartanburg, South Carolina

REFERENCES:
- [Background] Feenstra TL, van Genugten ML, Hoogenveen RT, Wouters EF, Rutten-van Molken MP. The impact of aging and smoking on the future burden of chronic obstructive pulmonary disease: a model analysis in the Netherlands. Am J Respir Crit Care Med. 2001 Aug 15;164(4):590-6. doi: 10.1164/ajrccm.164.4.2003167. PMID 11520721
- [Background] Ford ES, Croft JB, Mannino DM, Wheaton AG, Zhang X, Giles WH. COPD surveillance--United States, 1999-2011. Chest. 2013 Jul;144(1):284-305. doi: 10.1378/chest.13-0809. PMID 23619732
- [Background] Ford ES, Murphy LB, Khavjou O, Giles WH, Holt JB, Croft JB. Total and state-specific medical and absenteeism costs of COPD among adults aged >/= 18 years in the United States for 2010 and projections through 2020. Chest. 2015 Jan;147(1):31-45. doi: 10.1378/chest.14-0972. PMID 25058738
- [Background] Kern DM, Davis J, Williams SA, Tunceli O, Wu B, Hollis S, Strange C, Trudo F. Comparative effectiveness of budesonide/formoterol combination and fluticasone/salmeterol combination among chronic obstructive pulmonary disease patients new to controller treatment: a US administrative claims database study. Respir Res. 2015 Apr 23;16(1):52. doi: 10.1186/s12931-015-0210-x. PMID 25899176
- [Background] Mannino DM, Homa DM, Akinbami LJ, Ford ES, Redd SC. Chronic obstructive pulmonary disease surveillance--United States, 1971-2000. Respir Care. 2002 Oct;47(10):1184-99. PMID 12354338
- [Background] Murphy SL, Xu J, Kochanek KD. Deaths: final data for 2010. Natl Vital Stat Rep. 2013 May 8;61(4):1-117. PMID 24979972
- [Background] National Institutes of Health National Heart, Lung, and Blood Institute Fact Book Prevalence of Common Cardiovascular and Lung Diseases, U.S., 2007-2011. https://www nhlbi nih gov/about/documents/factbook/2012/chapter4 htm#4_5 ;2014.
- [Background] Simoni-Wastila L, Wei YJ, Qian J, Zuckerman IH, Stuart B, Shaffer T, Dalal AA, Bryant-Comstock L. Association of chronic obstructive pulmonary disease maintenance medication adherence with all-cause hospitalization and spending in a Medicare population. Am J Geriatr Pharmacother. 2012 Jun;10(3):201-10. doi: 10.1016/j.amjopharm.2012.04.002. Epub 2012 Apr 21. PMID 22521808
- [Background] van den Boom G, van Schayck CP, van Mollen MP, Tirimanna PR, den Otter JJ, van Grunsven PM, Buitendijk MJ, van Herwaarden CL, van Weel C. Active detection of chronic obstructive pulmonary disease and asthma in the general population. Results and economic consequences of the DIMCA program. Am J Respir Crit Care Med. 1998 Dec;158(6):1730-8. doi: 10.1164/ajrccm.158.6.9709003. PMID 9847260
- [Background] van der Molen T, Willemse BW, Schokker S, ten Hacken NH, Postma DS, Juniper EF. Development, validity and responsiveness of the Clinical COPD Questionnaire. Health Qual Life Outcomes. 2003 Apr 28;1:13. doi: 10.1186/1477-7525-1-13. PMID 12773199
- [Background] Simmons MS, Nides MA, Rand CS, Wise RA, Tashkin DP. Trends in compliance with bronchodilator inhaler use between follow-up visits in a clinical trial. Chest. 1996 Apr;109(4):963-8. doi: 10.1378/chest.109.4.963. PMID 8635378
- [Background] Clinical COPD Questionnaire website. http://ccq.nl/?page_id=15. Accessed January 15, 2016.
- See also: Clinical COPD Questionnaire website — http://ccq.nl/?page_id=15
- See also: D589CL00003_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4187&filename=D589CL00003_CSP_redacted.PDF
- See also: D589CL00003_SAP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4187&filename=D589CL00003_SAP_redacted.PDF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with chronic obstructive pulmonary disease (COPD) were recruited into 8 study sites in the United States from August 2016 to October 2017. The study evaluated the impact of medication reminders on adherence to Symbicort pressurized metered dose inhaler (pMDI) using a BreatheMate bluetooth device that monitored daily Symbicort inhaler use.
Pre-assignment Details: Subjects who entered the study already on a stable dose of Symbicort were enrolled and randomized at Visit 1 followed by a 26-week treatment period. Subjects who converted to Symbicort were enrolled at Visit 1 and entered a 25-day run-in period after which they were randomized at Visit 2, followed by a 26-week treatment period.
Groups:
- Control Group: All subjects took Symbicort pMDI budesonide/formoterol, 160/4.5 micrograms (mcg) x 2 actuations twice daily (BID), for oral inhalation from day 1 (baseline) of the treatment phase.
  Subjects randomized to the control group received Symbicort pMDI and a BreatheMate bluetooth monitoring device that monitored daily Symbicort inhaler use, as well as a study-supplied cellular phone that paired with the BreatheMate device to transmit data regarding Symbicort usage. Subjects in the control group did not receive any reminders to take their Symbicort or any feedback regarding medication compliance.
- Intervention Group: All subjects took Symbicort pMDI, budesonide/formoterol, 160/4.5 mcg x 2 actuations BID, for oral inhalation from day 1 (baseline) of the treatment phase.
  Subjects randomized to the intervention group received Symbicort pMDI, a BreatheMate bluetooth monitoring device that monitored daily Symbicort inhaler use, as well as a study-supplied cellular phone that paired with the BreatheMate device to transmit data regarding Symbicort usage. Subjects in the intervention group also received audio-visual daily reminders (beeps and flashes) to take their Symbicort on the BreatheMate Bluetooth monitoring device, and medication reminders from the cellular phone application.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 70 | 68
Full Analysis Set (FAS) (Subjects who took at least 1 inhalation of Symbicort during the treatment phase of the study.) | 70 | 67
Completed | 55 | 49
Not Completed | 15 | 19
Not completed — Eligibility Criteria Deviation | 2 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Device Technology Issue | 6 | 7
Not completed — Death | 0 | 1
Not completed — Did Not Start Treatment with Symbicort | 0 | 1
Not completed — Lost to Follow-up | 1 | 5
Not completed — Lost Device | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consisted of screened subjects who were randomized and took at least 1 inhalation of Symbicort during the treatment phase of the study (FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 70 | 67 | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (8.21) | 66.7 (8.72) | 66.7 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 60
  Male | 37 | 40 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 69 | 67 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 14 | 25
  White | 55 | 53 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Adherent Sets of Symbicort Puffs Per Day Over the 26-Week Study Period
Description: The mean number of adherent sets of Symbicort puffs per day for each group, over an average of 26 weeks was calculated. An adherent set of puffs was defined as exactly 2 sets of 2 Symbicort puffs per day. The 2 puffs that constitute a set must have been taken within 60 minutes of each other. A mean of 2.00 sets would be equal to 100% adherence (2 sets of 2 puffs). Subjects who did not take exactly 2 sets of 2 puffs on any given day throughout their device time on study were considered non-adherent for that day.
Time Frame: From baseline to end of treatment (EOT), (6 months).
Population: The FAS consisted of screened subjects who were randomized and took at least 1 inhalation of Symbicort during the treatment phase of the study.
Measure: Mean (Standard Deviation); unit: Adherent sets of puffs / day
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 70 | 67
Adherent sets of puffs / day | 1.3 (0.51) | 1.6 (0.39)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; The effect of medication reminders on Symbicort adherence was evaluated using a t-test. The equality of variances was also tested and as the variances were not equal, the Satterthwaite-t test was reported; Test type: Other; p < 0.001, Satterthwaite t-test

2. Secondary Outcome: Mean Clinical COPD Questionnaire (CCQ) Scores at Baseline, EOT, and Mean Change in Score Over the 26-Week Study Period.
Description: The CCQ is a 10-item measure of a subject's COPD symptoms, divided into 3 domains (Symptoms: Items 1, 2, 5 and 6; Functional State: Items 7, 8, 9, and 10; and Mental State: Items 3 and 4). Individual items within the CCQ were equally weighted. The total score was calculated by adding the scores of the 10 items and dividing that number by 10 (=number of items). In addition, individual domain scores were calculated. The total CCQ score and each of the 3 domain scores range from 0 (very good health status) to 6 (extremely poor health status). CCQ data was collected for all subjects at baseline and EOT visits. The mean CCQ total and domain scores at both baseline and 26 weeks (EOT) are presented along with the mean change from baseline at EOT or week 26. A positive change indicates worsening symptoms and a higher value is indicative of a poorer health status.
Time Frame: From baseline to EOT (6 months).
Population: The FAS consisted of screened subjects who were randomized and took at least 1 inhalation of Symbicort during the treatment phase of the study. Only subjects with CCQ results available for analysis are presented.
Measure: Mean (Standard Deviation); unit: Units on the CCQ scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 70 | 67
Units on the CCQ scale
  CCQ Total Score: Baseline: number analyzed (Participants) | 67 | 58
  CCQ Total Score: Baseline | 2.7 (0.97) | 2.2 (0.83)
  CCQ Total Score: EOT: number analyzed (Participants) | 67 | 58
  CCQ Total Score: EOT | 2.6 (1.08) | 2.4 (1.18)
  CCQ Total Score: Change from baseline: number analyzed (Participants) | 67 | 58
  CCQ Total Score: Change from baseline | -0.2 (0.99) | 0.2 (0.97)
  Symptom Score: Baseline: number analyzed (Participants) | 67 | 58
  Symptom Score: Baseline | 2.9 (1.07) | 2.4 (1.08)
  Symptom Score: EOT: number analyzed (Participants) | 67 | 58
  Symptom Score: EOT | 2.7 (1.11) | 2.4 (1.13)
  Symptom Score: Change from baseline: number analyzed (Participants) | 67 | 58
  Symptom Score: Change from baseline | -0.3 (1.13) | 0.0 (1.16)
  Functional State Score: Baseline: number analyzed (Participants) | 67 | 58
  Functional State Score: Baseline | 2.7 (1.39) | 2.2 (0.91)
  Functional State Score: EOT: number analyzed (Participants) | 67 | 58
  Functional State Score: EOT | 2.7 (1.36) | 2.6 (1.30)
  Functional State Score: Change from baseline: number analyzed (Participants) | 67 | 58
  Functional State Score: Change from baseline | 0.0 (1.32) | 0.4 (1.22)
  Mental State Score: Baseline: number analyzed (Participants) | 70 | 58
  Mental State Score: Baseline | 2.3 (1.37) | 1.6 (1.15)
  Mental State Score: EOT: number analyzed (Participants) | 67 | 67
  Mental State Score: EOT | 2.0 (1.42) | 1.7 (1.63)
  Mental State Score: Change from baseline: number analyzed (Participants) | 67 | 58
  Mental State Score: Change from baseline | -0.4 (1.50) | 0.2 (1.38)

3. Secondary Outcome: Mean Total and Domain Weekly CCQ Scores Over Each 2-Month Study Interval for the Intervention Group.
Description: The CCQ is a 10-item measure of a subject's COPD symptoms, divided into 3 domains (Symptoms: Items 1, 2, 5 and 6; Functional State: Items 7, 8, 9, and 10; and Mental State: Items 3 and 4). Individual items within the CCQ were equally weighted. The total score was calculated by adding the scores of the 10 items and dividing that number by 10 (=number of items). Individual domain scores were also calculated. The total CCQ score and each of the 3 domain scores range from 0 (very good health status) to 6 (extremely poor health status). Subjects in the intervention group took the CCQ weekly throughout the study. The 26-week treatment period was broken down into 3, 2-month intervals: Interval 1: from study day 1 to study day 63 (inclusive), Interval 2: study day 64 to study day 126 (inclusive), Interval 3: study day 127 to EOT (inclusive). The last week of each 2-month interval was used to represent that interval and results are presented for the total CCQ score and the 3 domain scores.
Time Frame: From baseline to EOT (6 months).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on the CCQ scale.
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
Units on the CCQ scale.
  CCQ Total Score: Interval 1, Week 9: number analyzed (Participants) | 39
  CCQ Total Score: Interval 1, Week 9 | 2.2 (1.06)
  CCQ Total Score: Interval 2, Week 18: number analyzed (Participants) | 35
  CCQ Total Score: Interval 2, Week 18 | 2.3 (1.07)
  CCQ Total Score: Interval 3, Week 27: number analyzed (Participants) | 2
  CCQ Total Score: Interval 3, Week 27 | 2.0 (0.14)
  CCQ Symptom Score: Interval 1, Week 9: number analyzed (Participants) | 39
  CCQ Symptom Score: Interval 1, Week 9 | 2.4 (1.24)
  CCQ Symptom Score: Interval 2, Week 18: number analyzed (Participants) | 35
  CCQ Symptom Score: Interval 2, Week 18 | 2.6 (1.26)
  CCQ Symptom Score: Interval 3, Week 27: number analyzed (Participants) | 2
  CCQ Symptom Score: Interval 3, Week 27 | 2.2 (0.23)
  CCQ Functional State Score: Interval 1, Week 9: number analyzed (Participants) | 39
  CCQ Functional State Score: Interval 1, Week 9 | 2.1 (1.09)
  CCQ Functional State Score: Interval 2, Week 18: number analyzed (Participants) | 35
  CCQ Functional State Score: Interval 2, Week 18 | 2.3 (1.09)
  CCQ Functional State Score: Interval 3, Week 27: number analyzed (Participants) | 2
  CCQ Functional State Score: Interval 3, Week 27 | 2.3 (0.47)
  CCQ Mental State Score: Interval 1, Week 9: number analyzed (Participants) | 39
  CCQ Mental State Score: Interval 1, Week 9 | 1.9 (1.25)
  CCQ Mental State Score: Interval 2, Week 18: number analyzed (Participants) | 35
  CCQ Mental State Score: Interval 2, Week 18 | 1.9 (1.28)
  CCQ Mental State Score: Interval 3, Week 27: number analyzed (Participants) | 2
  CCQ Mental State Score: Interval 3, Week 27 | 1.0 (0.71)

4. Secondary Outcome: Mean Number of Adherent Sets of Puffs Per Day for Each 2-Month Study Interval.
Description: The mean number of adherent sets of Symbicort puffs per day was calculated for each subject, for each of the 3, 2-month study intervals. Interval 1: from study day 1 to study day 63 (inclusive); Interval 2: study day 64 to study day 126 (inclusive); Interval 3: study day 127 to EOT (inclusive). A set is 2 puffs taken on the same calendar day, with the 2 puffs taken within 60 minutes of each other. The mean number of sets of Symbicort puffs per day was determined only for the days during device time on study for each subject.
Time Frame: From baseline to EOT (6 months).
Population: The FAS consisted of screened subjects who were randomized and took at least 1 inhalation of Symbicort during the treatment phase of the study. Only subjects with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: Adherent sets of puffs / day
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 70 | 67
Adherent sets of puffs / day
  Interval 1 | 1.4 (0.51) | 1.6 (0.37)
  Interval 2: number analyzed (Participants) | 68 | 65
  Interval 2 | 1.2 (0.61) | 1.6 (0.48)
  Interval 3: number analyzed (Participants) | 64 | 57
  Interval 3 | 1.2 (0.61) | 1.6 (0.51)

5. Secondary Outcome: Mean Number of Adherent Days Over the 26-Week Study Period.
Description: The total number of adherent days was defined as the number of treatment days a subject took 2 sets of 2 puffs of Symbicort and the inhalations in a puff set were within 60 minutes of each other. Subjects who did not take exactly 2 sets of 2 puffs on any given day throughout their device time on study were considered non-adherent for that day. The total number of adherent days for each subject was counted over the 26 week treatment period and the mean number of adherent days per group is presented.
Time Frame: From baseline to EOT (6 months).
Population: The FAS consists of screened subjects who were randomized and took at least 1 inhalation of Symbicort during the treatment phase of the study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 70 | 67
Days | 102.3 (50.76) | 128.4 (50.75)

6. Secondary Outcome: Mean Number of Symbicort Prescription Refills at Pharmacy Over the 26-Week Study Period.
Description: The total number of Symbicort prescriptions filled at a pharmacy during the 26-week treatment period was counted per subject. The mean number of Symbicort 30-day prescription refills per subject was then calculated and presented per group.
Time Frame: From baseline to EOT (6 months).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Number of Refills
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 70 | 67
Number of Refills | 5.1 (1.36) | 5.3 (1.29)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at the informed consent visit (Visit 1), at study day 90 and at the last follow-up telephone contact 30-days after the EOT visit on day 180 (approximately 7 months).
Groups:
- CONTROL GROUP: All subjects took Symbicort pMDI budesonide/formoterol, 160/4.5 mcg x 2 actuations BID, for oral inhalation from day 1 (baseline) of the treatment phase.
  Subjects randomized to the control group received Symbicort pMDI and a BreatheMate bluetooth monitoring device that monitored daily Symbicort inhaler use, as well as a study-supplied cellular phone that paired with the BreatheMate device to transmit data regarding Symbicort usage. Subjects in the control group did not receive any reminders to take their Symbicort or any feedback regarding medication compliance.
Arm/Group | CONTROL GROUP | INTERVENTION GROUP
All-Cause Mortality (participants affected / at risk) | 0/70 | 1/67
Serious Adverse Events (participants affected / at risk) | 5/70 | 8/67
Other Adverse Events (participants affected / at risk) | 18/70 | 15/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CONTROL GROUP (N=70) | INTERVENTION GROUP (N=67)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CONTROL GROUP (N=70) | INTERVENTION GROUP (N=67)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrolment was terminated early due to technical issues with the technologies provided at some clinical sites. The resulting impact on statistical power due to the reduced sample size likely imposes limits on the interpretability of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that within 2 years of study completion, the sponsor must review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT02864342/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02864342/SAP_001.pdf